CLINICAL TRIAL: NCT05283681
Title: A Phase 1 Study in Healthy Volunteers to Evaluate the Bioavailability of Risankizumab New Formulation in Pre-filled Syringe Relative to 90 mg/mL Formulation in Pre-filled Syringe and Characterization of Risankizumab Pharmacokinetics Using New Formulation in Auto-injector
Brief Title: A Study to Evaluate the Bioavailability of Risankizumab in Pre-filled Syringe or Auto-injector in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: M15-990
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — risankizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Risankizumab Dose A (Experimental): Participants will receive 1 Subcutaneous (SC) injection of risankizumab Dose A administered via Prefilled Syringe (PFS) at Day 1 and followed for 140 days
  Interventions: Drug: Risankizumab
- Risankizumab Dose B (Experimental): Participants will receive SC injections of risankizumab Dose B administered via PFS at Day 1 and followed for 140 days
  Interventions: Drug: Risankizumab
- Risankizumab Dose C (Experimental): Participants will receive 1 SC injection of risankizumab Dose C administered via Auto-Injector (AI) at Day 1 and followed for 140 days.
  Interventions: Drug: Risankizumab

INTERVENTIONS:
Drug: Risankizumab — Subcutaneous Injection via Prefilled Syringe (PFS)
  Other Names: ABBV-066; SKYRIZI
  Arms: Risankizumab Dose A; Risankizumab Dose B
Drug: Risankizumab — Subcutaneous Injection via Auto-Injector (AI)
  Other Names: ABBV-066; SKYRIZI
  Arms: Risankizumab Dose C

SUMMARY:
The objective of this study is to evaluate the bioavailability of risankizumab new formulation in prefilled syringe (PFS) relative to the 90 mg/mL formulation in PFS in healthy volunteers. The study will also evaluate the bioavailability of risankizumab new formulation in auto-injector (AI) relative to PFS in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male and female healthy volunteers between 18 and 55 years of age.
* Body weight less than 110.00 kg inclusive at Screening.

Exclusion Criteria:

* Previous exposure to any anti-IL-12/23 or anti-IL-23 treatment.
* Intention to perform strenuous exercise to which the subject is unaccustomed within one week prior to administration of study drug or during the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 226 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Up to 140 Days
  An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with the treatment. The investigator assesses the relationship of each event to the use of study drug.
Maximum observed serum concentration (Cmax) | Up to 113 Days
  Maximum observed serum concentration
Time to Cmax (Tmax) | Up to 113 Days
  Time to Cmax
Terminal phase elimination rate constant (β) | Up to 113 Days
  Terminal phase elimination rate constant
Terminal phase elimination half-life (t1/2) | Up to 113 Days
  Terminal phase elimination half-life
Area under the concentration-time curve (AUC) from time 0 to time of the last measurable concentration (AUCt) | Up to 113 Days
  AUC from 0 to time of last measurable concentration
AUC from time 0 to infinity (AUCinf) | Up to 113 Days
  AUC from time 0 to infinity
Number of Anti-drug antibody (ADA) Titers | Up to 113 Days
  Incidence of anti-drug antibodies

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (2):
- United States (2):
  - Acpru /Id# 210844, Grayslake, Illinois
  - PPD Clinical Research Unit - Austin /ID# 211456, Austin, Texas

IPD SHARING:
Plan to Share IPD: No